CLINICAL TRIAL: NCT06232421
Title: A Prospective, Parallel, Single-blind Clinical Study Using Stratified Randomization of the Effectiveness, Tolerability and Safety of the Medicinal Product "Foscelantan, Medicinal Plate 4.0x5.0 cm in Package No. 1" Produced by UNITEKHPROM BSU, Republic of Belarus, in Comparison With the Medicinal Product Povidone- Iodine Produced by BelAseptika JSC, in Adult Patients With Purulent-inflammatory Processes of the Skin and Soft Tissues Due to the Neuropathic Form of Diabetic Foot Syndrome or Chronic Venous Insufficiency, Phase I-II of the Wound Process
Brief Title: Clinical Study in Adult Patients With Purulent-inflammatory Processes of the Skin and Soft Tissues, Phase I-II of the Wound Process
Acronym: OLENKRON-01
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Research Institute for Physical Chemical Problems of the Belarusian State University (Other)
Collaborators: Vitebsk Regional Clinical Hospital (Other Government); Unitary Enterprise UNITEHPROM BSU (Unknown); The 10th Minsk City Clinical Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OLENKRON-01
Record Dates: First submitted 2024-01-07; First posted 2024-01-30 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Foot Infections; Chronic Venous Insufficiency
Keywords: diabetic foot infection; chronic venous insuffiency; lidocaine; cellulose; miramistin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients with the neuropathic form. Treatment with Foscelantan (Experimental): A prospective, parallel, single-blind clinical study using stratified randomization of the effectiveness, tolerability and safety of the drug "Foscelantan, medicinal plate 4.0×5.0 cm in package No. 1" produced by UNITEHPROM BSU, Republic of Belarusin adult patients with purulent-inflammatory processes of the skin and soft tissues due to the neuropathic form of diabetic foot syndrome, phase I-II wound process. All patients will receive systemic traditional therapy for the underlying and concomitant diseases.
  Interventions: Drug: Foscelantan
- Patients with the neuropathic form. Treatment with Povidone-iodine (Active Comparator): A prospective, parallel, single-blind clinical study using stratified randomization of the effectiveness, tolerability and safety of the drug Povidone-iodine produced by BelAseptika JSC, in adult patients with purulent-inflammatory processes of the skin and soft tissues due to the neuropathic form of diabetic foot syndrome, phase I-II wound process. All patients will receive systemic traditional therapy for the underlying and concomitant diseases.
  Interventions: Drug: Povidon-iodine
- Patients with chronic venous insufficiency. Treatment with Foscelantan (Experimental): A prospective, parallel, single-blind clinical study using stratified randomization of the effectiveness, tolerability and safety of the drug "Foscelantan, medicinal plate 4.0×5.0 cm in package No. 1" produced by UNITEHPROM BSU, Republic of Belarus in adult patients with purulent inflammatory processes of the skin and soft tissues due to chronic venous insufficiency," phase I-II of the wound process. All patients will receive systemic traditional therapy for the underlying and concomitant diseases.
  Interventions: Drug: Foscelantan
- Patients with chronic venous insufficiency. Treatment with Povidone-iodine (Active Comparator): A prospective, parallel, single-blind clinical study using stratified randomization of the effectiveness, tolerability and safety of the drug Povidone-iodine produced by BelAseptika JSC, in adult patients with purulent-inflammatory processes of the skin and soft tissues due to chronic venous insufficiency", phase I-II of the wound process . All patients will receive systemic traditional therapy for the underlying and concomitant diseases.
  Interventions: Drug: Povidon-iodine

INTERVENTIONS:
Drug: Foscelantan — "Foscelantan, medicinal plate 4.0x5.0 cm in package No. 1" produced by UNITEHPROM BSU, Republic of Belarus
  Arms: Patients with chronic venous insufficiency. Treatment with Foscelantan; Patients with the neuropathic form. Treatment with Foscelantan
Drug: Povidon-iodine — Povidone-iodine solution 100 mg/ml produced by BelAseptika CJSC, Republic of Belarus
  Arms: Patients with chronic venous insufficiency. Treatment with Povidone-iodine; Patients with the neuropathic form. Treatment with Povidone-iodine

SUMMARY:
The purpose of this study is to estimate efficiency, tolerance, safety of "Foscelantan, medicinal plate 4.0x5.0 cm in package No. 1" among adult patients who have purulent-inflammatory processes of the skin and soft tissues due to the neuropathic form of diabetic foot syndrome or chronic venous insufficiency, phase I-II of the wound process.

DETAILED DESCRIPTION:
Diabetes takes the third place in the World in terms of its medical and social significance. Diabetes is often complicated with such urulent-inflammatory processe as diabetic foot syndrome. Urulent-inflammatory processes treatment takes a long time and medications due to microcirculation disorders, metabolic disorders, progressive hypoxia and a number of other factors. A moist wound environment, conducive to the natural process of wound cleansing (autolysis), regeneration of damaged tissue, and reduction of pain, irreversible sorption of excess exudate and toxic components and easy removal of the drug from the surface of the wound without additional trauma or damage are yhe main conditions of successful wound healing.Wound dressings made of fibrous polysaccharides modyfied with drugs meet these requirements. Foscelantan has prolonged antimicrobial, analgesic and reparative action, has the ability to transform on the wound surface into an amorphous gel-like mass, irreversibly bind wound detritus and pathological exudate, and provide optimal conditions for the process of wound healing.

ELIGIBILITY:
Inclusion Criteria:

* The presence of purulent-inflammatory processes of the skin and soft tissues due to the neuropathic form of diabetic foot syndrome (Main diagnosis: Diabetes mellitus type I or II, clinical metabolic compensation/subcompensation, class I - II according to the Wagner classification) or chronic venous insufficiency (Main diagnosis: Varicose veins dilatation of the veins of the lower extremities, class C6 according to the CEAP classification), phase I-II of the wound process
* The size of the ulcerative defect is from 1 cm² to 20 cm²
* Secondary type of wound healing
* Absence of exposed bones and tendons in the wound
* Absence of severe concomitant diseases in the stage of decompensation, oncological diseases, as well as diseases requiring steroid therapy
* Availability of written informed consent from the patient to participate in the study
* The patient's ability to follow the instructions of the research physician and comply with the study regimen

Exclusion Criteria:

* Individual intolerance or hypersensitivity reactions to the components of the drug Foscelantan
* Neuroischemic form of diabetic foot syndrome
* The presence of serious concomitant pathology (severe form of renal and hepatic failure, systemic connective tissue diseases, severe cardiovascular insufficiency), history and current mental illness
* The need to constantly take drugs from the list of prohibited therapies
* Participation of the patient in another clinical trial within 3 months before the current clinical trial
* Acute bleeding
* Level of peripheral blood leukocytes less than 1.5 × 109 per l, platelets less than 75.0 × 109 per l.
* Hemoglobin less than 80g per l.
* Positive tests for syphilis, human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Severe liver dysfunction - AST or ALT levels exceed the upper limit of normal by 5 times or more, bilirubin ≥ 2.0 mg/dL (34.2 µmol/L).
* Severe renal dysfunction - creatinine 2 times higher than reference values
* Diabetes mellitus in a state of clinical and metabolic decompensation
* Pregnant and breastfeeding women
* At one's own request without explaining the reasons for the action.
* At the request of the research physician, if the research subject violates the protocol requirements for diet, consumption of alcoholic beverages, and medications without the prescription of the research physician.
* For reasons independent of the study subject and the research physician, when a study subject develops drug intolerance and other life-threatening or requiring emergency pharmacotherapy adverse reactions to the administration of the study drug.
* The need to prescribe drugs from the list of prohibited treatments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with trophic ulcers cured | 15 days
  Number of patients cured

SECONDARY OUTCOMES:
percentage reduction in the non-epithelialized area of the wound surface in relation to the initial one | 15 days
  Additionally, the percentage reduction in the non-epithelialized area of the wound surface relative to the original will be calculated, determined by digital non-contact planimetry during dressing changes. This indicator will be assessed using a digital camera and image analysis software

CONTACTS AND LOCATIONS:
Locations (2):
- Belarus (2):
  - 10th CITY CLINICAL HOSPITAL, Minsk, Minsk City
  - Health care institution Vitebsk Regional Clinical Hospital, Vitebsk, Vitebsk Oblast

IPD SHARING:
Plan to Share IPD: No